CLINICAL TRIAL: NCT04047030
Title: The Mobility Toolkit: Electronically Augmented Assessment of Functional Recovery Following Lower-extremity Trauma
Acronym: MBTK
Status: Completed | Type: Observational
Sponsor: Major Extremity Trauma Research Consortium (Other)
Responsible Party: Sponsor
Other Study IDs: W81XWH-18-1-0815
Record Dates: First submitted 2019-07-26; First posted 2019-08-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Gait

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Injured Cohort: Approximately 300 participants treated for a fracture of the tibial plateau, pilon, ankle or calcaneus will be enrolled from METRC civilian trauma centers and military treatment facilities over an 18 month period. Participating centers treat large numbers of severe orthopaedic injuries and have a proven track record for successfully recruiting and retaining participants in prospective studies in orthopaedic trauma. Participants will be enrolled following definitive treatment of their injury.
  Interventions: Other: None- Observational Study
- Non-Injured Volunteers: Non-injured adults of similar age and gender distribution will be enrolled at two participating centers (Carolinas Medical Center and Womack Military Medical Center). The sample of non-injured volunteers will exclude individuals with history of lower extremity injury, vascular disease, or who require use of ambulatory aides to walk.
  Interventions: Other: None- Observational Study

INTERVENTIONS:
Other: None- Observational Study — No Intervention

SUMMARY:
The study will prospectively enroll and follow 300 participants ages 18-60 surgically treated for a lower-extremity articular injury including fractures of the tibial plateau, pilon, ankle, and calcaneus.

DETAILED DESCRIPTION:
The study will prospectively enroll and follow 300 participants ages 18-60 surgically treated for a lower-extremity articular injury including fractures of the tibial plateau, pilon, ankle, and calcaneus. All participating centers will undergo training to implement the Mobility Toolkit (MTK). Research Staff will facilitate a series of performance tests while participants wear the MTK device. MTK assessment will also be conducted on 150 non-injured adults matched to the injured cohort on age and gender. These individuals will be enrolled and assessed once at two participating centers. Study flow and data capture are summarized in the figure on the next page.

ELIGIBILITY:
Inclusion Criteria:

1. 18-60 years of age
2. Open or closed fractures of the tibial plateau, pilon, ankle or calcaneus requiring surgical fixation.

Exclusion Criteria:

1. Gustilo type IIIB or IIIC injuries
2. No other surgically or non-surgically treated injuries that impact gait (e.g. upper extremity injury proximal to the elbow; spinal cord injury; contralateral or ipsilateral fractures).
3. Neurologic impairment or deficit that impairs gait
4. Prior injuries or conditions that alter gait (e.g. severe osteoarthritis)
5. Severe problems with maintaining follow-up (e.g. participants who are prisoners, who are intellectually challenged without adequate family support, or have documented psychiatric disorders).
6. Unable to provide informed consent in English or Spanish.

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Adults ages 18-60 surgically treated for a fracture of the tibial plateau, pilon, ankle, or calcaneus at one of 10 participating centers. Patients meeting the inclusion and exclusion criteria will approached for enrollment in to the study.
Sampling Method: Non-Probability Sample
Enrollment: 244 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Ease of use of the Mobility Toolkit during clinic | 12 months
  Feasibility will be assessed through surveys of study participants and clinical staff to document time and burden of using MTK during clinic visits.
Satisfaction of the Mobility Toolkit | 12 months
  Satisfaction will be assessed through surveys of study participants and clinical staff to document time and burden of using MTK during clinic visits.
Gait Quality assessed with Mobility Tooklkit | 12 months
  Gait Quality will be measured using the MTK to assess gait parameters such as lift acceleration, step time asymmetry, and peak-to-peak upper body pitch and roll.
Gait Quality assessed by performance tests | Change in gate from measured at 3, 6 & 12 months
  Gait will be assessed while completing three performance tests: 10 meter walk, sit to stand, and timed up and go (TUG) Injured participants will be assessed at time of first weight bearing, and at clinic visits 3, 6 and 12 months following definitive treatment.
Physical Function | Change in physical function measured at 3, 6, & 12 months
  Patient Reported Function will be assessed using the physical function item banks from the Patient Reported Outcomes Measurement Information System (PROMIS). Injured participants will be assessed at baseline and at each follow-up visit.
Pain Score | Change in pain score measured at 3, 6, & 12 months
  Patient Reported Pain will be assessed using the pain interference item banks from the Patient Reported Outcomes Measurement Information System (PROMIS). Injured participants will be assessed at baseline and at each follow-up visit.
Number of patient complications resulting from injury | 12 months
  Injury related complications such as infection, non-union, and hardware failure will be captured prospectively the year following treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Sims, MD, Principal Investigator — Carolinas Medical Center; Lisa Reider, PhD, Principal Investigator — JHSPH/METRC
Locations (10):
- United States (10):
  - University of Kentucky, Lexington, Kentucky
  - University of Maryland R Adams Cowley Shock Trauma Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Barnes Jewish Hospital, St Louis, Missouri
  - Mission Hospital, Asheville, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Womack Army Medical Center at Ft. Bragg, Fort Bragg, North Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Health Science Center - Houston, Houston, Texas
  - San Antonio Military Medical Center (SAMMC), San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Data sharing beyond manuscripts and scientific presentations will be processed through the METRC website in the short term. Currently, a standard form will be available for researchers outside METRC to request access to final data generated from METRC studies. These requests will be transmitted to the METRC Coordinating Center for initial review to make sure the relevant materials are provided in support of the request. METRC is committed to making data as widely available as possible while safeguarding the privacy of study participants and protecting the intellectual property of the Consortium.
  Data will only be made available after it is completely stripped of identifiable information such as dates, geographic locators, and any other event information which is sufficiently rare as to make it possible to deduce the identity of an individual participant. When necessary for complete de-identification, data may be grouped.